CLINICAL TRIAL: NCT04706598
Title: A Phase I/II Single Arm Study of Intravesical Administration With Camrelizumab for High-risk Non-muscle Invasive Bladder Cancer(NMIBC) Failing in BCG Treatment
Brief Title: Safety and Efficacy of Camrelizumab for High-risk NMIBC Failing BCG Treatment
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Shen Kang Hospital Development Center (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-UC-II-004
Record Dates: First submitted 2020-12-27; First posted 2021-01-13 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Urinary Bladder Neoplasms; Immunotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravesical therapy group (Experimental): Camrelizumab(SHR-1210) is administered on the first day of each treatment cycle (D1) at a dose up to 200 mg. The recommended phase II dose(RP2D) to be decided after safety run-in.
  The cycle is divided into an induction course and a maintenance course. The induction course is initiated 2 weeks after TURBT and repeat once a week for 6 weeks . After that, the maintenance course starts every 3 weeks. The maximum duration of dosing is 2 years.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Solution for Infusion (Intravesical)
  Other Names: SHR-1210

SUMMARY:
This study will evaluate the safety and efficacy of bladder intravesical Camrelizumab in patients with high-risk non-muscle-invasive bladder cancer who failed BCG therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically-confirmed diagnosis of high risk non-muscle-invasive urothelial cell carcinoma of the bladder (mixed histology tumors allowed if urothelial carcinoma histology is >50%).
3. Fully resected disease at study entry (residual CIS acceptable).
4. BCG-unresponsive high risk non-muscle-invasive bladder cancer after treatment with adequate BCG therapy(at least five times a week during the induction phase and at least two times a week during the maintenance phase).
5. Ineligible for radical cystectomy or refusal of radical cystectomy.
6. Consent to tissue specimen retrieval and testing.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Adequate normal organ and marrow function as defined below:

   1. Haemoglobin (HB) ≥ 90 g/L
   2. Absolute neutrophil count (ANC) ≥1.5×10^9/L(no granulocyte colony-stimulating factor support for 2 weeks before day 1 of cycle 1)
   3. Lymphocyte count≥0.500×10^9/L
   4. Platelet count ≥100×10^9/L(No blood transfusions within 2 weeks before day 1 of cycle 1)
   5. 4.0×10^9/L≤White Blood Cell Count (WBC)≤15×10^9/L
   6. AST (SGOT)/ALT (SGPT)/Alkaline phosphatase ≤ 2.5 x institutional upper limit of normal(ULN) (excluded Gilbert's disease patients, whose serum bilirubin level ≤ 3x ULN)
   7. INR/aPTT≤1.5×ULN(Which only applies to patients not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be given a stable dose)
   8. Serum creatinine (Cr) ≤ 1.5 times the upper institutional limit of normal (ULN) or Serum creatinine Cl>60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976)
9. Women of childbearing potential who have a negative serum pregnancy test within 72 hours prior to the first dose should consent to and must use effective contraception during and for 6 months after the end of the study.
10. Men should consent to patients who must use contraception during the study and for 6 months after the end of the study period.
11. The subject is personally willing and able to provide written informed consent to be able to comply with the protocol.

Exclusion Criteria:

1. Muscle-invasive, locally advanced nonresectable, or metastatic urothelial carcinoma.
2. Concurrent extra-vesical (i.e., urethra, ureter, or renal pelvis)urothelial cell carcinoma.
3. Have participated in a clinical trial of an investigational drug or device within 4 weeks prior to receiving the first treatment in this project.
4. Received chemotherapy, targeted small molecule therapy, immunotherapy or radiation therapy following a recent cystoscopy or transurethral resection of a bladder tumour.
5. History of other malignancies within the last 5 years.
6. Active autoimmune disease that has required systemic treatment in the past 2 years.
7. History of idiopathic pulmonary fibrosis (including pneumonia), drug-induced pneumonia, histoplasmosis (i.e. occlusive bronchiolitis, cryptogenic histoplasmosis), or evidence of active pneumonia on chest CT scan (history of fibrosis in radiation pneumonia), patients with active tuberculosis.
8. Active infection requiring systemic therapy,therapeutic oral or intravenous (IV) antibiotics within 14 days prior to enrolment (patients receiving prophylactic antibiotics (e.g. for the prevention of urinary tract infections or chronic obstructive pulmonary disease) can be enrolled).
9. Patients who are pregnant or breastfeeding, or expecting to conceive .
10. Previous treatment with anti-PD-1 monoclonal antibody, PD-L1 monoclonal antibody, CTLA-4 monoclonal antibody, or other drugs that act on T-cell co-stimulation or any other antibody of the checkpoint pathway.
11. Patients with known positive test for human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS).
12. Patients with known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (Hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU/ml; Hepatitis C reference: HCV antibody positive and HCV viral copy number > upper limit of normal value).
13. Received a live virus vaccine within 30 days of planned start of study treatment.
14. Has had an allogeneic tissue/solid organ transplant.
15. Long-term oral steroids, more than 10 mg/day of methandrostenolone or similar, must be stopped for 28 days before entry into the group.
16. Evidence of apparently uncontrolled concomitant disease that may affect compliance with the protocol or interpretation of the results, including significant liver disease (e.g. cirrhosis, uncontrolled major seizures or superior vena cava syndrome).
17. Significant cardiovascular disease, such as New York Heart Association heart attack (class II or higher), myocardial infarction, unstable arrhythmia or unstable angina within 3 months prior to study entry.
18. Patients who have had major surgery within 4 weeks prior to study entry, or who are expected to require major surgery during the course of the study, except diagnostic procedures such as TURBT or biopsy.
19. History of autoimmune diseases, including but not limited to severe muscle weakness, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, angio-thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, dry syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
20. History of severe allergy, sensitisation or other hypersensitivity reactions to chimeric or humanised antibodies or fusion proteins.
21. Patients who, in the opinion of the investigator, are otherwise unable to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The maximum dose of Camrelizumab for intravesical treatment | 3 months after trial initiation(Phase I)
  The maximum tolerated dose (MTD) of Camrelizumab that will be given intravesically to patients with BCG-refractory NMIBC(de-escalated doses of 200/150/100mg) and recommended for phase II studies (RP2D).
Event-Free Survival (EFS) | 3 months after patient treatment (Phase II)
  Recurrence of high-grade cancer (TaHG, T1HG, CIS), or disease progression to stage T2 or beyond or lymph node metastasis or distant metastasis, or the need for other treatment (including systemic chemotherapy, radical cystectomy, radiation therapy), and death from any cause.

SECONDARY OUTCOMES:
Incidence of adverse events | Until progressive disease or death
  Incidence of adverse events and treatment-related adverse events
Assessment of HGRF | 6 months and 1 year after patient enrollment
  High grade cancer recurrence free rate (HGFR) at 6 months and 1 year of treatment.
Assessment of RFS | 6 months and 1 year after patient enrollment
  Recurrence free survival (RFS) at 6 months and 1 year of treatment.
Assessment of PFS | 6 months and 1 year after patient enrollment
  Progression free survival (PFS) at 6 months and 1 year of treatment.
the predictive value of PD-1 expresssion | 1 year after patient enrollment
  the predictive value of PD-L1 expression assessed in tumor tissue and urine sample obtained before and after Camrelizumab instillation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Wang, MD, Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Yushan Liu, MD, Study Director — Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine; Xudong Yao, MD, Study Director — Shanghai Tenth People's Hospital,Shanghai Tong Ji University School of Medicine
Locations (4):
- China (4):
  - Shanghai Ninth People's Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital,Shanghai Tong Ji University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sylvester RJ, Oosterlinck W, van der Meijden AP. A single immediate postoperative instillation of chemotherapy decreases the risk of recurrence in patients with stage Ta T1 bladder cancer: a meta-analysis of published results of randomized clinical trials. J Urol. 2004 Jun;171(6 Pt 1):2186-90, quiz 2435. doi: 10.1097/01.ju.0000125486.92260.b2. PMID 15126782
- [Result] Taniguchi K, Koga S, Nishikido M, Yamashita S, Sakuragi T, Kanetake H, Saito Y. Systemic immune response after intravesical instillation of bacille Calmette-Guerin (BCG) for superficial bladder cancer. Clin Exp Immunol. 1999 Jan;115(1):131-5. doi: 10.1046/j.1365-2249.1999.00756.x. PMID 9933432
- [Result] Mitropoulos DN. Novel insights into the mechanism of action of intravesical immunomodulators. In Vivo. 2005 May-Jun;19(3):611-21. PMID 15875784
- [Result] Kamat AM, Flaig TW, Grossman HB, Konety B, Lamm D, O'Donnell MA, Uchio E, Efstathiou JA, Taylor JA 3rd. Expert consensus document: Consensus statement on best practice management regarding the use of intravesical immunotherapy with BCG for bladder cancer. Nat Rev Urol. 2015 Apr;12(4):225-35. doi: 10.1038/nrurol.2015.58. Epub 2015 Mar 24. PMID 25800393
- [Result] Witjes JA, Palou J, Soloway M, Lamm D, Kamat AM, Brausi M, Persad R, Buckley R, Colombel M, Bohle A. Current clinical practice gaps in the treatment of intermediate- and high-risk non-muscle-invasive bladder cancer (NMIBC) with emphasis on the use of bacillus Calmette-Guerin (BCG): results of an international individual patient data survey (IPDS). BJU Int. 2013 Oct;112(6):742-50. doi: 10.1111/bju.12012. Epub 2013 Mar 1. PMID 23452187
- [Result] Oddens JR, Sylvester RJ, Brausi MA, Kirkels WJ, van de Beek C, van Andel G, de Reijke TM, Prescott S, Witjes JA, Oosterlinck W. The effect of age on the efficacy of maintenance bacillus Calmette-Guerin relative to maintenance epirubicin in patients with stage Ta T1 urothelial bladder cancer: results from EORTC genito-urinary group study 30911. Eur Urol. 2014 Oct;66(4):694-701. doi: 10.1016/j.eururo.2014.05.033. Epub 2014 Jun 16. PMID 24948466
- [Result] Chang SS, Bochner BH, Chou R, Dreicer R, Kamat AM, Lerner SP, Lotan Y, Meeks JJ, Michalski JM, Morgan TM, Quale DZ, Rosenberg JE, Zietman AL, Holzbeierlein JM. Treatment of Nonmetastatic Muscle-Invasive Bladder Cancer: American Urological Association/American Society of Clinical Oncology/American Society for Radiation Oncology/Society of Urologic Oncology Clinical Practice Guideline Summary. J Oncol Pract. 2017 Sep;13(9):621-625. doi: 10.1200/JOP.2017.024919. Epub 2017 Aug 10. No abstract available. PMID 28796558
- [Result] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Result] Dinney CP, Greenberg RE, Steinberg GD. Intravesical valrubicin in patients with bladder carcinoma in situ and contraindication to or failure after bacillus Calmette-Guerin. Urol Oncol. 2013 Nov;31(8):1635-42. doi: 10.1016/j.urolonc.2012.04.010. Epub 2012 May 9. PMID 22575238
- [Result] Couzin-Frankel J. Breakthrough of the year 2013. Cancer immunotherapy. Science. 2013 Dec 20;342(6165):1432-3. doi: 10.1126/science.342.6165.1432. No abstract available. PMID 24357284
- [Result] Inamura K. Bladder Cancer: New Insights into Its Molecular Pathology. Cancers (Basel). 2018 Apr 1;10(4):100. doi: 10.3390/cancers10040100. PMID 29614760
- [Result] Catalona WJ, Hudson MA, Gillen DP, Andriole GL, Ratliff TL. Risks and benefits of repeated courses of intravesical bacillus Calmette-Guerin therapy for superficial bladder cancer. J Urol. 1987 Feb;137(2):220-4. doi: 10.1016/s0022-5347(17)43959-0. PMID 3806806
- [Result] Pietzak EJ, Bagrodia A, Cha EK, Drill EN, Iyer G, Isharwal S, Ostrovnaya I, Baez P, Li Q, Berger MF, Zehir A, Schultz N, Rosenberg JE, Bajorin DF, Dalbagni G, Al-Ahmadie H, Solit DB, Bochner BH. Next-generation Sequencing of Nonmuscle Invasive Bladder Cancer Reveals Potential Biomarkers and Rational Therapeutic Targets. Eur Urol. 2017 Dec;72(6):952-959. doi: 10.1016/j.eururo.2017.05.032. Epub 2017 Jun 3. PMID 28583311
- [Result] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Result] Zhu J, Armstrong AJ, Friedlander TW, Kim W, Pal SK, George DJ, Zhang T. Biomarkers of immunotherapy in urothelial and renal cell carcinoma: PD-L1, tumor mutational burden, and beyond. J Immunother Cancer. 2018 Jan 25;6(1):4. doi: 10.1186/s40425-018-0314-1. PMID 29368638
- [Result] Inman BA, Sebo TJ, Frigola X, Dong H, Bergstralh EJ, Frank I, Fradet Y, Lacombe L, Kwon ED. PD-L1 (B7-H1) expression by urothelial carcinoma of the bladder and BCG-induced granulomata: associations with localized stage progression. Cancer. 2007 Apr 15;109(8):1499-505. doi: 10.1002/cncr.22588. PMID 17340590
- [Result] He YT, Li DJ, Liang D, Zheng RS, Zhang SW, Zeng HM, Chen WQ, He J. [Incidence and mortality of bladder cancer in China, 2014]. Zhonghua Zhong Liu Za Zhi. 2018 Sep 23;40(9):647-652. doi: 10.3760/cma.j.issn.0253-3766.2018.09.002. Chinese. PMID 30293387